CLINICAL TRIAL: NCT00662506
Title: A Phase Ib/II Study of AZD2171 in Combination With Daily Temozolomide and Radiation in Patients With Newly Diagnosed Glioblastoma Not Taking Enzyme-Inducing Anti-epileptic Drugs
Brief Title: Cediranib, Temozolomide, and Radiation Therapy in Treating Patients With Newly Diagnosed Glioblastoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00267; NCI-2009-00267 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MGH-07-344; PHS 398/2590; CDR0000593717; PHS 398/2590 (Other: Massachusetts General Hospital Cancer Center); 8030 (Other: CTEP); P30CA006516 (NIH); R01CA129371 (NIH)
Record Dates: First submitted 2008-04-18; First posted 2008-04-21 (Estimated); Last update posted 2023-06-06 (Actual); Status verified 2017-09

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — cediranib; Diffusion Tensor Imaging; Fluorodeoxyglucose F18; Radiotherapy, Intensity-Modulated; Magnetic Resonance Spectroscopy; Temozolomide

ARMS (1):
- Treatment (enzyme inhibitor therapy, chemotherapy, IMRT) (Experimental): See Detailed Description
  Interventions: Drug: Cediranib Maleate; Procedure: Diffusion Tensor Imaging; Procedure: Diffusion Weighted Imaging; Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging; Radiation: Fludeoxyglucose F-18; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Procedure: Perfusion Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Drug: Temozolomide

INTERVENTIONS:
Drug: Cediranib Maleate — Given PO
  Other Names: AZD2171; AZD2171 Maleate; Recentin
Procedure: Diffusion Tensor Imaging — Undergo DTI
  Other Names: DTI
Procedure: Diffusion Weighted Imaging — Undergo T1 weighted DCE-MRI
  Other Names: Diffusion Weighted MRI; Diffusion-Weighted Magnetic Resonance Imaging; Diffusion-Weighted MR Imaging; Diffusion-Weighted MRI; DWI; DWI MRI; DWI-MRI; MR Diffusion-Weighted Imaging
Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging — Undergo DCE-MRI
  Other Names: DCE MRI; DCE-MRI; DYNAMIC CONTRAST ENHANCED MRI
Radiation: Fludeoxyglucose F-18 — Undergo 18 FDG PET
  Other Names: 18FDG; FDG; fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Perfusion Magnetic Resonance Imaging — Undergo PWI
  Other Names: magnetic resonance perfusion imaging
Procedure: Positron Emission Tomography — Undergo 18 F FDG-PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET SCAN; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac

SUMMARY:
This phase I/II trial is studying the side effects and best dose of cediranib to see how well it works when given together with temozolomide and radiation therapy in treating patients with newly diagnosed glioblastoma. Cediranib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving cediranib together with temozolomide and radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety profile and optimal dose of AZD2171 (cediranib) (15mg or 20mg or 30mg) in combination with temozolomide and radiation in patients with newly diagnosed glioblastoma (Phase Ib) II. To determine median progression-free survival of patients with newly diagnosed glioblastoma treated with AZD2171 in combination with temozolomide and radiation (Phase II)

SECONDARY OBJECTIVES:

I. To determine the radiographic response proportion in newly diagnosed glioblastoma patients with measurable disease. (Phase II) II. To determine the median overall survival. (Phase II) III. To determine the "vascular normalization" window in newly diagnosed glioblastoma patients by the application of serial, non-invasive, MRI parameters. (Phase II) IV. To measure the glucose metabolism changes in a subset of newly diagnosed glioblastoma patients by performing FDG PET studies. (Phase II) V. Measurement of circulating endothelial and progenitor cells and plasma levels of VEGF-A; VEGF-B; VEGF-C; VEGF-D; sVEGFR1, sVEGFR2, bFGF, PlGF, PDGF-AA; PDGF-AB; PDGF-BB; SDF1α; tumstatin; thrombospondin-1; interleukin-8; collagen IV sICAM1, sVCAM1 as markers for response to AZD2171 in newly diagnosed glioblastoma patients. (Phase II) VI. Correlation of treatment outcomes with pre-AZD2171 tumor specimens with respect to cell proliferation, apoptosis, microvascular density (MVD), basement membrane and pericyte coverage, angiopoietin-1 and -2 expression to determine whether these immunohistochemical analyses can be predictive of the response to AZD2171. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of cediranib followed by a phase II study.

Patients begin study treatment within 21-42 days after craniotomy or 14-21 days after stereotactic biopsy.

PHASE Ib:

CHEMORADIOTHERAPY: Patients receive cediranib orally (PO) once daily and oral temozolomide once daily for 6 weeks. Within 2-6 hours of dosing, patients undergo concurrent intensity-modulated radiotherapy (IMRT) once daily, 5 days a week for 6 weeks. Cediranib monotherapy: Patients receive cediranib PO once daily for 4 weeks (weeks 7-10). Cediranib and temozolomide monthly therapy: Patients receive cediranib PO once daily for 24 weeks (weeks 11-34) and temozolomide once daily, 5 days a week in weeks 11, 15, 19, 23, 27, and 31. Cediranib monotherapy: Patients receive a fixed-dose of cediranib once daily for 24 weeks (weeks 35-58).

PHASE II:

CHEMORADIOTHERAPY: Patients receive cediranib PO at the recommended phase II dose determined in phase Ib, temozolomide PO, and undergo concurrent IMRT as in phase Ib (weeks 1-6). Cediranib monotherapy: Patients receive cediranib PO (at the recommended phase II dose determined in phase Ib) once daily for 4 weeks (weeks 7-10). Cediranib and temozolomide monthly therapy: Patients receive cediranib PO (at the recommended phase II dose determined in phase Ib) once daily for 24 weeks (weeks 11-34) and temozolomide once daily, 5 days a week in weeks 11, 15, 19, 23, 27, and 31. Cediranib monotherapy: Patients receive a fixed-dose of cediranib once daily for 24 weeks (weeks 35-58).

Patients undergo blood and urine sample collection at baseline and periodically during study. Blood samples are measured for tumstatin, as well as other well established biomarkers, including VEGF-A, -D, sVEGFR1, sVEGFR2, sICAM1, sVCAM1, PlGF, PDGF-AA, PDGF-AB, PDGF-BB, thrombospondin-1, and IL-8 by electrochemiluminescence detection. Circulating endothelial cell (CEC) assays are evaluated to assess the kinetics of CECs and progenitor cells prior to and during antiangiogenic therapy with cediranib and chemoradiotherapy. Urine samples are collected for proteomic analyses to evaluate serial change of growth factors such as VEGF and PlGF and of matrix metalloproteinases in response to treatment with cediranib. Archival tumor tissue is collected for analysis of tumor microvascular density, basement membrane and pericyte coverage, angiopoietin-1 and -2 expression, tumor cell proliferation, and apoptosis by immunostaining methods and immunoenzyme techniques.

Patients also undergo dynamic contrast enhanced (DCE)-MRI and T2-weighted or perfusion-weighted MRI at baseline and periodically during study to monitor antiangiogenic effect on tumor vasculature through parameters reflecting both tumor perfusion and permeability; and diffusion tensor imaging to measure degree of water diffusion and fractional anisotropy. A subset of patients undergo fludeoxyglucose F 18 positron emission tomography (FDG-PET) periodically to monitor antiangiogenic effects on glucose utilization.

After completion of study treatment, patients are followed periodically for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed glioblastoma

  * Newly diagnosed disease
* Scheduled to receive standard post-surgical (i.e., biopsy or resection) temozolomide and radiotherapy
* Must have residual, contrast-enhancing tumor (≥ 1 centimeter in ≥ 1 dimension)
* Patients must be maintained on a stable corticosteroid regimen for 5 days prior to their baseline scan and for 5 days prior to their first vascular MRI; the dose of steroids should remain the same during the baseline vascular MRIs
* Archival tumor tissue available for molecular analysis
* No intratumoral hemorrhage or peritumoral hemorrhage by MRI
* Karnofsky performance status 60-100%
* Leukocytes ≥ 3,000/mcl
* Absolute neutrophil count ≥ 1,500/mcL
* Platelet count ≥ 100,000/mcL
* Hemoglobin ≥ 8 g/dL
* Total bilirubin normal
* AST/ALT ≤ 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Proteinuria ≤ 1+ on two consecutive dipsticks ≥ 7 days apart
* Mini-mental status examination score ≥ 15
* Must be able to tolerate MRI and must consent to participate in additional Vascular Imaging Procedures per protocol

  * CT scans cannot be substituted for MRI
* Mean QTc ≤ 500 msec (with Bazett's correction) by electrocardiogram
* No concurrent malignancy except curatively treated basal cell or squamous cell carcinoma skin cancer or carcinoma in situ of the cervix or breast

  * Patients with prior malignancies must be disease-free for ≥ 5 years
* No history of familial long QT syndrome or other significant ECG abnormality
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to cediranib
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Hypertension (e.g., blood pressure > 140/90 mm Hg)
  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would preclude study compliance
* No known coagulopathy that increases risk of bleeding
* No history of clinically significant hemorrhages in the past
* No New York Heart Association class III-IV heart disease
* No condition requiring concurrent drugs or biologics with proarrhythmic potential
* No other concurrent chemotherapy agents, investigational agents, or biologic therapy
* No prior chemotherapy, radiotherapy, or any experimental therapy for this disease
* No prior IV bevacizumab for any other medical condition
* No prior carmustine implant (Gliadel Wafer)
* No prior brachytherapy or radiosurgery for this disease
* More than 30 days since prior and no other concurrent investigational agents or participation in an investigational therapeutic trial
* At least 2 weeks since prior and no concurrent enzyme-inducing anti-epileptic drugs (EIAEDs)

  * Concurrent non-EIAEDs allowed
* No concurrent CYP450-inducing anticonvulsants
* No concurrent anticoagulants (e.g., dalteparin, warfarin, or low-molecular weight heparin)

  * If patients require warfarin or other anticoagulants (e.g., low-molecular weight heparin) while on study, then patient may continue treatment
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent VEGF inhibitors
* No concurrent pentamidine
* No concurrent herbal or nontraditional medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (Phase II) | At day 218
  The fraction of patients alive and free of disease progression after the MRI scan scheduled. This fraction will be compared, using a one sample, two-sided exact binomial test, to 50% progression-free survival (PFS). For safety assessment, the study will be powered to ensure at least 85% chance of observing a serious adverse event, if the probability of such an event on treatment were >=5%.
Safety profile and optimal dose of cediranib during chemoradiotherapy (Phase I) | Up to 30 days after the last dose
  A dose-limiting toxicity of cediranib is defined as a clinically significant adverse event or abnormal laboratory value assessed as unrelated to disease progression, intercurrent illness, or concomitant medications/temozolomide and occurs following the first dose of cediranib in the chemoradiation.

SECONDARY OUTCOMES:
Blood biomarkers (Phase II) | Up to 1 year
  Log-transformation is expected to yield approximately homogenous and symmetric standard errors, both for Poisson events and quantities obtained by assays with successive dilutions. We will plot the median levels and quartiles over time. First, we will compare on-study values to baseline, than we will test for an association between treatment time and markers, using a linear mixed effects model with log-transformed data and a spline function of time. The two-sided, paired t-test test will be powered to detect an effect-size of 0.5.
MRI parameters (Phase II) | Up to 48 weeks
  The comparisons of all MRI measurements will be against their day -1 values (baseline), using a 2-sided, paired Wilcoxon test (Hollander and Wolfe 1973).
Tumor biomarkers (Phase II) | At baseline
  Exploratory analyses will be performed to determine if there is any correlation between the molecular/vascular phenotype of the tumor or quantitative measurements, we will use for this purpose ANOVA on log-transformed marker measurements. We will analyze changes in the measurements, and correlate biomarkers with clinical and radiographic response, similarly as for blood and urine biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth R Gerstner, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Hoebel KV, Bridge CP, Ahmed S, Akintola O, Chung C, Huang RY, Johnson JM, Kim A, Ly KI, Chang K, Patel J, Pinho M, Batchelor TT, Rosen BR, Gerstner ER, Kalpathy-Cramer J. Expert-centered Evaluation of Deep Learning Algorithms for Brain Tumor Segmentation. Radiol Artif Intell. 2024 Jan;6(1):e220231. doi: 10.1148/ryai.220231. PMID 38197800
- [Derived] Hoebel KV, Patel JB, Beers AL, Chang K, Singh P, Brown JM, Pinho MC, Batchelor TT, Gerstner ER, Rosen BR, Kalpathy-Cramer J. Radiomics Repeatability Pitfalls in a Scan-Rescan MRI Study of Glioblastoma. Radiol Artif Intell. 2020 Dec 16;3(1):e190199. doi: 10.1148/ryai.2020190199. eCollection 2021 Jan. PMID 33842889
- [Derived] Emblem KE, Farrar CT, Gerstner ER, Batchelor TT, Borra RJ, Rosen BR, Sorensen AG, Jain RK. Vessel caliber--a potential MRI biomarker of tumour response in clinical trials. Nat Rev Clin Oncol. 2014 Oct;11(10):566-84. doi: 10.1038/nrclinonc.2014.126. Epub 2014 Aug 12. PMID 25113840
- [Derived] Pinho MC, Polaskova P, Kalpathy-Cramer J, Jennings D, Emblem KE, Jain RK, Rosen BR, Wen PY, Sorensen AG, Batchelor TT, Gerstner ER. Low incidence of pseudoprogression by imaging in newly diagnosed glioblastoma patients treated with cediranib in combination with chemoradiation. Oncologist. 2014 Jan;19(1):75-81. doi: 10.1634/theoncologist.2013-0101. Epub 2013 Dec 5. PMID 24309981